CLINICAL TRIAL: NCT00011661
Title: Social Network Based Intervention to Reduce Lead Exposure Among Native American Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 8755-CP-001
Record Dates: First submitted 2001-02-26; First posted 2001-02-28 (Estimated); Last update posted 2006-09-04 (Estimated); Status verified 2006-09

CONDITIONS: Lead Poisoning
Keywords: Lead poisoning; Native Americans
MeSH Terms: conditions — Lead Poisoning

INTERVENTIONS:
Behavioral: Education on behaviors to reduce lead exposure

SUMMARY:
The purpose of this study is to examine whether adding an inter-generational component to an existing social network-based lay health advisor intervention increases its effectiveness in mobilizing a Native American community to respond to heavy metal contamination from lead and zinc mining.

DETAILED DESCRIPTION:
Ottawa County, Oklahoma, the site of the research, was heavily mined for zinc and lead in the first half of this century. Mine tailings containing heavy metals are stored in large piles up to 200 feet in height. Ottawa County is home to 8 Indian tribes and much of the mine waste is on tribal land. Specifically, the study will: a) integrate existing Native American youth programs with the existing lay health advisor intervention (Society of Clan Mothers and Fathers) to form an inter-generational intervention, b) expand the existing lay health advisor intervention to address cadmium in addition to lead, c) use participatory research methods to involve tribal youth and adults in an air monitoring study, d) assess the extent to which the intervention contributes to belief, attitude and behavior changes that will reduce heavy metal exposure and absorption in Native American children; and e) assess the contribution of the intervention to creating changes in organizational, community, tribal and government (city, county, state, federal) capacity to address heavy metal contamination in Ottawa County, Oklahoma.

ELIGIBILITY:
Children ages 1-6

Live in Ottawa County, Oklahoma

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400
Dates: Start 2000-06; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Locations (1):
- Wyandotte Nation, Wyandotte, Oklahoma, United States